CLINICAL TRIAL: NCT05127330
Title: Pilot RCT of a Video-based Intervention for Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504431
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Suicidal Ideation; Suicidal Behaviors; Suicide
Keywords: Psychiatric Hospitalization
MeSH Terms: conditions — Suicidal Ideation; Suicide | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LifePlans (Experimental): LifePlans is a video series using real patients telling their stories of overcoming suicidal thoughts and behaviors to help others who are struggling with these issues.
  Interventions: Behavioral: LifePlans
- Treatment as Usual (Active Comparator): Individuals will receive unrestricted routine care only.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: LifePlans — LifePlans is a video-based intervention, in which patients watch episodes starting during a psychiatric hospitalization and continuing through 1 month post-discharge. Other mental health treatment is unrestricted.
  Arms: LifePlans
Behavioral: Treatment as Usual — Individuals will receive unrestricted routine mental health care in the community as appropriate for their condition.
  Arms: Treatment as Usual

SUMMARY:
The investigators will develop a brief video-based intervention for suicide prevention, called LifePlans. LifePlans will be tested in a pilot randomized controlled trial (n = 40) to examine its feasibility and acceptability. Investigators will recruit patients admitted to a psychiatric hospital for suicidal thoughts and behaviors who will receive the intervention for 4 weeks post-discharge. Patients will be assessed at hospital baseline, 1 month post-discharge, and 6 months post-discharge.

DETAILED DESCRIPTION:
In this project, we propose to develop a new intervention, called LifePlans. LifePlans will consist of brief videos that highlight patients' experiences. Episodes will cover these topics: 1) developing a personalized "Life Plan" to stay safe and restrict means, 2) clarifying valued life domains and related goals to improve hopefulness, 3) using informal problem solving to cope better with illness, 4) improving communication with family/friends to increase social support, and 5) adhering to primary treatments including pharmacotherapy and psychotherapy to promote illness management. LifePlans will be tested in a pilot randomized controlled trial (n = 40) to examine its feasibility and acceptability. Investigators will recruit patients admitted to a psychiatric hospital for suicidal thoughts and behaviors who will receive the intervention for 4 weeks post-discharge. Patients will be assessed at hospital baseline, 1 month post-discharge, and 6 months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* current psychiatric hospitalization for suicidal thoughts and behaviors
* 18 years or older
* ability to speak and read English
* access to means for viewing videos (computer, tablet, smartphone)

Exclusion Criteria:

* current psychotic symptoms
* current cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital; Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Upload to NIMH Data Archive
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after the completion of the study and stored permanently.
Access Criteria: Refer to NIMH Data Archive for details.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 92 participants were approached for the study, and 40 were consented and enrolled in the study after it was determined that they met eligibility criteria.
Period: Overall Study
Arm/Group | LifePlans | Treatment as Usual
Started | 19 | 21
Completed | 10 | 14
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LifePlans | Treatment as Usual | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (12.8) | 40.0 (15.9) | 36.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 18 | 16 | 34
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 19 | 21 | 40
Columbia Suicide Severity Rating Scale (C-SSRS) [Mean (Standard Deviation); unit: score on scale] — The Columbia Suicide Severity Rating Scale is an interviewer-rated measure of suicidal thoughts and behaviors. The total score (sum of items) will be used and ranges from 2 to 25 with higher scores indicating higher suicidal thoughts and behaviors.
  score on scale | 14.5 (2.6) | 13.6 (2.7) | 14.0 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The Client Satisfaction Questionnaire is a self-report measure of patient satisfaction with treatment. The total score will be used and ranges from 8 to 32 with increased scores indicating greater satisfaction with treatment.
Time Frame: 1 Month
Population: Difference due to missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LifePlans | Treatment as Usual
Number analyzed (Participants) | 7 | 14
score on scale | 25.6 (3.1) | 24.6 (14)

2. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia Suicide Severity Rating Scale is an interviewer-rated measure of suicidal thoughts and behaviors. The total score (sum of items) will be used and ranges from 2 to 25 with higher scores indicating higher suicidal thoughts and behaviors.
Time Frame: 1 Month
Population: Difference due to missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LifePlans | Treatment as Usual
Number analyzed (Participants) | 10 | 14
score on scale | 7.6 (6.9) | 6.1 (5.1)

ADVERSE EVENTS:
Time Frame: 1 Month
Arm/Group | LifePlans | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/14
Other Adverse Events (participants affected / at risk) | 0/10 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifePlans (N=10) | Treatment as Usual (N=14)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This is a treatment development study and therefore was not designed to test the efficacy of the intervention given the small sample size. Instead, the goal was to examine feasibility and acceptability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT05127330/Prot_SAP_000.pdf